CLINICAL TRIAL: NCT05261074
Title: Impact of COVID-19 Confinement on Foreign Body Ingestion in the Pediatric Emergency Department
Brief Title: Foreign Body Ingestion During COVID-19 Lockdown
Acronym: COCE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP-COCE
Record Dates: First submitted 2022-02-28; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Foreign Body Ingestion
Keywords: Foreign body; Children; Covid-19; Oesophagus
MeSH Terms: conditions — Foreign Bodies; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention (retrospective study)

SUMMARY:
Ingestion of foreign bodies (FB) is one of the most observed domestic accidents and a frequent reason for consultation in pediatric emergency departments (PED). In the United States, nearly 100,000 ingestions of FB have been recorded by the National Poison Data System (NPDS), which represented the 4th cause of intoxication in 2015.

Ingestion of FB involves very different mechanisms in children and adult patients. Unlike adults, 98% of FB ingestions in children are accidental and involve common objects found at home environment. Ingested FBs are of many types and vary depending on the object composition of the child's environment and supervision. The lockdown for COVID-19 pandemic highly modified children environment and parent supervision. Children remained at home and parents lived at home for teleworking.

In this study, the modifications of children environment that could affect epidemiology of FB ingestion will be evaluated. This is a retrospective study with a sample of around > 100 children of Louis Mourier hospital from January 1 to December 31, 2019 and from March 1 to May 31, 2020. The total duration of the study is planned for 10 months.

Primary outcomes:

• To determine the role of COVID-19 pandemic linked containment on the prevalence of FB ingestions in children.

Secondary outcomes:

* Describe the epidemiological-clinical, radiological, therapeutic and evolutionary characteristics of the FB consultant's ingestions in the emergency department
* Determine the frequency of endoscopy or surgery
* Determine the factors favoring the use of endoscopic extraction From March 16 to May 10, 2020.

DETAILED DESCRIPTION:
To analyze the impact of COVID-19 lockdown in 2020 on FB ingestion by children, to compare epidemiology of FB ingestion during 3 periods: 2020 lockdown (March to May 2020), the entire 2019 year and March to May 2019. The anonymized data will be entered in Epidata software and data transfer secured using APHP servers.

The variables of interest will include: sex, age at the time of ingestion, type of the FB, single or multiple ingestion, annual period of ingestion, ingestion schedule, existence of a witness, time of arrival at the emergency room, presence and nature of clinical symptoms of ingestion, position of the FB in the digestive tract, complications of this ingestion, x-ray exams used to locate FB need for an extraction gesture, nature of this gesture, completion time, successes and complications of extraction.

The population should have an estimated number of between 100-150 children. Descriptive statistics. The quantitative variables will be described as mean and standard deviation or as median, quartiles, minimum and maximum depending on whether their distribution is Gaussian or not. The qualitative variables will be described in numbers (percentage).

Comparison tests. Qualitative data will be analyzed using Chi2 or Fischer's exact test.

The study was approved by hospital's ethics committee.

ELIGIBILITY:
Inclusion Criteria:

* Children <15 years old.
* Child who consulted in the pediatric emergency department of Louis-Mourier University Hospital.
* For ingestion of foreign bodies coded in Urqual software.

Exclusion Criteria:

* Refusal to participate in the study
* unusable files (> 20% missing data out of a total of 40 major items),
* Ingestion of CE was suspected but not confirmed,
* Ingestion of caustics or other chemicals,
* Introduced from an FB into the digestive tract by a route other than the oral cavity.

Ages: 1 Day to 15 Years | Sex: All
Age Groups: Child
Study Population: Child who consulted in the pediatric emergency department of Louis-Mourier University Hospital for ingestion of foreign bodies coded in Urqual software.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-10-20 (Estimated); Study Completion 2022-10-20 (Estimated)

PRIMARY OUTCOMES:
Prevalence of foreign body (FB) ingestions in children | 1 year
  To determine the role of COVID-19 pandemic linked containment on the prevalence of foreign body (FB) ingestions in children

CONTACTS AND LOCATIONS:
Overall Officials: Jerôme VIALA, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Louis Mourier Hospital - Assistance Publique Hopitaux de Paris, Colombes, France

IPD SHARING:
Plan to Share IPD: No